CLINICAL TRIAL: NCT06680427
Title: Siegel™ Transcatheter Aortic Valve Replacement System (TAVR) Early Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MiRus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR-001
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis Symptomatic
Keywords: Transcatheter Aortic Valve Replacement; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Device: Siegel Transcatheter Aortic Valve (TAVR)

INTERVENTIONS:
Device: Siegel Transcatheter Aortic Valve (TAVR) — Replacement of native aortic valve with the Siegel Transcatheter Aortic Valve (TAVR) by a transfemoral approach.

SUMMARY:
The Siegel™ Transcatheter Aortic Valve (TAVR) early feasibility study objective is to assess the acute and long-term safety and feasibility of the Siegel TAVR device in adult subjects with symptomatic, severe native aortic stenosis eligible for the transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
The Siegel™ Transcatheter Aortic Valve (TAVR) Early Feasibility Study is a prospective, non-randomized, single-arm, multi-center study conducted in the US. The primary objective is to assess the acute and long-term safety and feasibility of the Siegel TAVR device in adult subjects with symptomatic, severe native aortic stenosis eligible for the transcatheter aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for entry in this study if all the following conditions are met:

1. Symptomatic, severe native aortic stenosis in subjects 50 years or older Aortic Valve Area (AVA) ≤ 1.0 cm2 or Aortic Valve Area (AVA) index ≤ 0.6 cm2/m2 and Jet velocity ≥ 4.0 m/s or mean gradient ≥ 40 mmHg or dimensionless Index <0.25
2. New York Heart Association Functional Class ≥ 2
3. Requires aortic valve replacement and is indicated for TAVR as determined by the Heart Team (composed of an experienced interventional cardiologist and an experienced cardiac surgeon)
4. Eligible for transfemoral delivery of the Siegel TAVR
5. Native aortic annulus suitable for safe placement of Siegel 23mm or 26mm transcatheter heart valve (preprocedural measurements by Transthoracic Echocardiogram (TTE) and Computed Tomography (CT) of area derived aortic annulus diameter)
6. Understands the study requirements and the treatment procedures and provides written informed consent
7. Subject agrees to complete all required scheduled follow-up visits.

Exclusion Criteria:

Subjects will be excluded for entry in this study if any of the following conditions are met:

Anatomical

1. Anatomy precluding safe placement of Siegel TAVR
2. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
3. Pre-existing prosthetic heart valve in any position (note, mitral ring is not an exclusion).
4. Unicuspid or bicuspid aortic valve
5. Severe aortic regurgitation (>3+)
6. Severe mitral or severe tricuspid regurgitation(>3+) requiring intervention.
7. Moderate to severe mitral stenosis.
8. Hypertrophic obstructive cardiomyopathy
9. Echocardiographic evidence of intracardiac mass, thrombus or vegetation requiring treatment.
10. Severe basal septal hypertrophy with outflow gradient Clinical
11. Evidence of an acute myocardial infarction ≤ 30 days before enrollment.
12. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the index procedure
13. Blood dyscrasias as defined: leukopenia (WBC < 3000 cell/mL, anemia (Hgb < 9 g/dL), thrombocytopenia (platelet count < 50,000 cells/mL), history of bleeding diathesis or coagulopathy.
14. Untreated clinically significant Coronary Artery Disease (CAD) requiring revascularization
15. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support within the past 30 days.
16. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of enrollment
17. Need for emergency surgery for any reason
18. Ventricular dysfunction with left ventricular ejection fraction (LVEF) < 30% as measured by resting echocardiogram
19. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
20. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of enrollment
21. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy, or end stage renal disease requiring chronic dialysis
22. GI bleeding within the past 3 months
23. Severe lung disease with Forced Expiratory Volume in 1 second (FEV1) < 50% predicted or currently on home oxygen
24. History of cirrhosis or any active liver disease
25. Significant frailty as determined by the Heart Team (after objective assessment of frailty parameters).
26. Significant abdominal or thoracic aortic disease (such as porcelain aorta, abdominal aortic aneurysm > 5.0 cm, severe calcification, aortic coarctation, etc.) that would preclude safe passage of the delivery system or cannulation and aortotomy for surgical AVR .
27. Severe pulmonary hypertension (e.g., pulmonary artery systolic pressure ≥ 2/3 systemic pressure)
28. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin, heparin, molybdenum, rhenium, ticlopidine and clopidogrel, contrast media
29. Ongoing sepsis, including active endocarditis
30. Body Mass Index (BMI) > 50 kg/m2
31. Subject refuses a blood transfusion
32. Life expectancy < 24 months due to associated non-cardiac co-morbid conditions
33. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent
34. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
35. Currently participating in an investigational drug or another investigational device trial
36. Subject is contraindicated for cardiac computed tomography (CT).
37. Subject belongs to a vulnerable population (Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Technical success of implantation of the Siegel TAVR | Immediate post procedure
  Technical success will be reported as freedom from mortality, successful device implant, and freedom from surgery or intervention related to the device.
All-cause mortality or disabling stroke | 30 Days
  Mortality will be reported as rate of death/mortality at 30 days. Disabling stroke will be reported according to Valve Academic Research Consortium (VARC-3) Guidelines

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford, Palo Alto, California
  - NCH Healthcare System, Naples, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - Columbia University Medical Center/ NYPH, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided